CLINICAL TRIAL: NCT05014542
Title: Needling Techniques for Tonifying Kidneys and Dredging Meridians for Knee Osteoarthritis: A Randomized Clinical Trial
Brief Title: Needling Techniques for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Svijetlana Perculija Durdevic (Other)
Collaborators: Nanjing University of Chinese Medicine, Xueping Zhou, Li Ren (Unknown); School of Medicine, University of Zagreb, Pero Hrabac (Unknown); Health Center Zagreb East, Ljiljana Karadakic (Unknown)
Responsible Party: Sponsor-Investigator, Svijetlana Perculija Durdevic, Head of Family Medicine Practice, Principal Investigator, Family Medicine Practice Svijetlana Perculija Durdevic, MD
Organization: Family Medicine Practice Svijetlana Perculija Durdevic, MD (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39603233785
Record Dates: First submitted 2021-08-08; First posted 2021-08-20 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis; Kidney Yin Deficiency; Kidney Yang Deficiency
Keywords: Needling; Techniques; Randomized; Reinforcing; Reducing; Acupuncture
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy; Analgesics

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, interventional, prospective.
Who Masked: Outcomes Assessor
Masking Description: The assessor of the physiatrists' measures and the assessor in charge of helping fill in WOMAC, VAS, KDSQ, DRUG, and Lequesne index were blind to the fact to which group participants belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Experimental): Participants in Acupuncture group will get acupuncture treatments to their symptomatic knee/knees according to the study protocol. Acupuncture will be provided to participants in three cycles, each three weeks duration, with frequency three times weekly. Period between the cycles is three weeks long. Participants will get acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) which dose could vary according to participant symptoms intensity. Participants and investigator are not blinded for treatment type.
  Interventions: Procedure: Acupuncture; Drug: Conventional Medical Treatment
- Control Group (Active Comparator): Participants in Control group will get their standard conventional treatment (analgesics) which dose could vary according to participant symptoms intensity. Participants and investigator are not blinded for treatment type.
  Interventions: Drug: Conventional Medical Treatment

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment is 30 minutes. All treatments will be equal.
  Arms: Acupuncture Group
Drug: Conventional Medical Treatment — Participants could take their standard conventional medical treatment or analgesics. Analgesics therapy is prescribed by their general practitioner. The dose of analgesics could be modified according to participants' symptoms intensity.
  Other Names: Analgesics

SUMMARY:
The thirty-nine-week open-label clinical study investigates the efficacy of acupuncture for Knee Osteoarthritis (KOA) as adjunctive therapy to analgesics compared to analgesics only and assesses the effects after 9 and 24 weeks, with safety assessment provided.

The study seeks to find possible additional benefits of acupuncture on Kidney Deficiency (KD) while treating KOA with an acupuncture protocol designed to treat KOA following Traditional Chinese Medicine (TCM) theory, which connects KOA with KD as its root cause. The points prescription uses local and Kidney-related points to treat KOA.

The chronic conditions require a higher number of acupuncture treatments. This study will provide acupuncture treatments in three cycles, each three weeks long, with frequency three times weekly. Twenty-seven acupuncture treatments of KOA during fifteen weeks tend to improve KOA and KDS; symptoms are assessed in 10 successive time points, and treatment effects and effect persistence are analysed.

64 patients with symptomatic KOA are randomly allocated into the Acupuncture (A) or Control (C) group according to their permanent, unique, and coincidental Personal Identification Number, which is randomly given to all citizens in Croatia. Before the experiment starts, demographics and disease parameters of all participants are compared. To objectify acupuncture effects, the enrolled physiatrist's measures included knee measures at 3 time points: baseline, at the end of acupuncture (Week 15), and nine weeks later (Week 24). Subjective evaluations of symptoms are assessed by Western Ontario and McMaster University Arthritis Index (WOMAC) total and subscales scores, Numeric Rating Scale (NRS), and Kidney Deficiency Syndrome Questionnaire (KDSQ) every 3 weeks till the 24th week (9 assessments). Analgesics taken by participants (DRUG) in the last three days before the assessments are recorded. Acupuncture treatment was promised to all participants. Therefore, at Week 25, the between-group analysis ended, and the C group crossed over to receive the identical acupuncture protocol. The 10th assessment in Week 39 was used to estimate, by within-group analysis, the immediate effects of the acupuncture in group C and the effect persistence in group A.

The Lequesne index was introduced additionally at Week 24 as another measure of the knee's functional state.

DETAILED DESCRIPTION:
KOA's high prevalence assures the trial's participation motivation of patients regarding associated pain and functional impairment. Besides pain and stiffness, patients experience muscle weakness, poor balance, and joint distortion in an advanced stage. KOA attacks the diseased ones at the age of 50. Pain worsens with joint loading and becomes relieved by rest. KOA supposes bones remodelling, cartilage thinning, synovial thickening, and joint space narrowing. The advanced stage is presented by joint instability, squaring, and even subluxation.

KOA involves both knees and the contributing symptoms of old age from the scope of Kidney deficiency syndromes, such as weakness, insomnia, depression, tinnitus, forgetfulness, feeling cold, hot, low back pain, thirst at night, and disturbed urination could be manifested.

The acupuncture treatment of KOA follows syndrome differentiation. The treatment principle distinguishes the deficient root (primary Kidney deficiency and secondary Blood deficiency) as the cause, and the excessive branch (knee bone Bi syndrome) when in empty Cou Li spaces, the external factor becomes entraped, consequently. An aspiration with treatment is to tonify the Kidney, nourish Qi, tonify and invigorate Blood, remove Damp and Cold by transferring them toward the deficiency rather than expelling, and relieve the channels and collaterals from the obstruction. Moreover, knee meridians should be dredged to improve knee symptoms by a simultaneous reinforcing-reducing technique on local points and reinforcing on KD-related points. Eventually, the improvements of KD indicate better life quality.

The study's design involves two groups: an acupuncture (A) group that receives acupuncture treatment adjunctive to analgesics, and a control (C) group that receives only analgesics. Participants were recruited from the target population of patients over 50 from 2 Family Medicine practices with confirmed KOA. The study sample was formed with inclusion and exclusion criteria. 64 patients were recruited. All medical data of the participants were available to the investigator. After fulfilling the SOAP form (Subjective, Objective, Assessment, Plan) and getting informed written consent, the study sample was randomly allocated into two groups by size of their permanent, unique eleven-digit long Personal Identification Numbers (OIB), which is assigned to all Croatian citizens. Its first ten digits are accidentally chosen, and the last is a control number. Every second participant ordered by the size of OIB belongs to the same group; odd ones belong to the A group, and even ones to the C group. Demographic and disease parameters are compared at baseline to determine if the groups are comparable. All study participants received analgesics and could modify dosages according to their needs. Analgesics were nonsteroidal anti-inflammatory drugs (NSAIDs) and/or tramadol. Taken analgesics were recorded at Weeks 0, 3, 6, 9, 12, 15, 18, 21, 24, and 39. The dose represents an average daily dose of analgesics from the last three days. The dose was recorded after conversion to the comparable dose of the selected representative (ibuprofen), the most prescribed one. The given data will be statistically processed and analyzed.

Patients in the A group started with acupuncture treatment in September 2021, with the first treatment cycle. Each of the 3 treatment cycles, in total, is three weeks long, each consists of 9 treatments, patients will receive acupuncture three times per week and the two adjacent acupuncture cycles are separated by three weeks without acupuncture.

Acupuncture treatment protocol includes local treatment points Dubi (ST-35), Neixiyan (EX-LE-4) and Heding (EX-LE-2), Xuehai (SP-10), Yanglingquan (GB-34), Yinlingquan (SP-9), Zusanli (ST-36), Sanyinjiao (SP-6), and points targeting Kidney deficiency syndrome Taixi (KI-3), Guanyuan (CV 4), and Shenshu (BL-23).

Disposable sterile acupuncture needles 0.30 × 40 mm are used. The depth and angle procedure predicted straight needling on 1-1.5 inches deep, with a mild reinforcing-reducing method for local points, further straight and 0.5-1 inch deep with the reinforcing method for points based on KD syndromes. Complete treatment lasts 30 minutes, and the manipulations are provided every 10 minutes, three times in total.

The sample size was calculated based on the Berman et al. (1999) study. The sample size was calculated by envisioning a two-sided test with unequal variances: type I error 0,05, power 0,95. Group sample sizes of 16 and 16 (i.e. complete study population of 32 subjects) achieve 95,78% power to reject the null hypothesis of equal means and with a significance level (alpha) of 0,050 using a two-sided two-sample unequal-variance t-test.

From a longer treatment period of this study and higher participants' drop-off expected, the population was doubled to 64 subjects in total.

Research methods were determined upon the clinical question "Could the prolonged design of acupuncture treatments on patients with knee osteoarthritis (KOA) decrease pain and improve the function of the knee joints and additionally achieve positive effects on the debilitating symptoms of a Kidney deficiency as a root cause of KOA, measured by recognized questionnaires?".

Evaluation of the therapeutic effects of acupuncture on KOA included WOMAC, VAS, KDSQ scores, and DRUG at Weeks 0, 3, 6, 9, 12, 15, 18, 21, 24, and 39. WOMAC is a renowned questionnaire for KOA evaluation. It measures 5 items for pain, 2 for stiffness, and 17 for functional limitation. VAS is a continuous numeric rating scale of 100 mm in length that is widely used for pain intensity assessment. The KDSQ questionnaire is a valid and reliable measure constructed in 2012 to evaluate Kidney Yin and Yang deficiency syndromes of Hong Kong Chinese middle-aged women by Chen et al. KDSQ represents a valid questionnaire for KD assessment in this study population.

From a total of 10 assessments, the first 9 compared scores between groups A and C. Participants were promised to receive equal acupuncture treatment if they were randomised into the C group. So, group C crossed over to receive the identical protocol from Week 25 to 39, and the 10th assessment was added to both groups of participants to estimate the immediate effects of the acupuncture treatment in the C group and estimate treatment effect persistence in the A group over 24 weeks, in a within-group manner. The physiatrist's assessments at 3 time-points (baseline, 15th Week, and 24th Week) include the standard physiatrist KOA measurements (knee and thigh circumference, range of motion of the knee). The Lequesne index was added as the knee's functional state measure in Week 24.

Data is stored electronically with secured and restricted access. Data transfer will be encrypted, and all data that could identify individuals has been removed.

Study analysis serves to process the effects of acupuncture treatment. Baseline data are obtained before the experiment starts. Besides immediate effects, effects persistence was assessed at Weeks 24 (9 weeks after acupuncture of group A ended) and 39. WOMAC total score at the end of the acupuncture protocol (Week 15) is a primary outcome, while WOMAC subscales, VAS, and KDSQ scores, DRUG at Weeks 15, 24 and 39, and persistence of WOMAC total were secondary and supportive of the primary one. Secondary outcome measures include physiatrists' measures and the Lequesne index as well. Effect sizes are calculated from data comparison to the control group up to Week 24 or baseline at Week 39. Analyses were performed on 64 participants, randomised for the intention-to-treat (ITT) analysis using the maximum available data set (i.e. excluding the missing values) from repeated measures of variables of interest and their variances. ITT analysis, excluding missing values, was selected regarding dropouts that emerged in the study, completely random without any causal clustering. Dropouts produced missing values. Omitting missing values can compromise the statistics and produce bias. Therefore, sensitivity analyses were provided to compare those who dropped out and those who completed the study to determine if data significantly differed. Also, a test calculation with the Last observation carried forward technique (LOCF) with the imputed last observed value in the missing one was performed to check if the obtained effects still stand. All statistical tests are two-sided. The Shapiro-Wilk test tests the normality distribution. The non-parametric Mann-Whitney U test was used for comparability testing with 95% power and α=0,05. The main efficacy indicators tested the comparability of the groups with the Mann-Whitney U test and quantified observed effects by mean differences and Cohen's d.

A participant will be considered to have withdrawn from the trial when consent is revoked or if the participant cannot be contacted or located. Participants will not be withdrawn from the trial for protocol violations. Withdrawal due to an adverse event should be distinguished from withdrawal due to insufficient response.

All adverse events will be recorded in the Adverse Event Report Form at every treatment. If this happens, an adverse event will be followed until its resolution. The serious adverse event must be reported to the Medical Ethics Committee.

It is expected to relieve pain and increase joint mobility, along with alleviating KD and reducing the use of analgesics and confirming the safety of acupuncture.

This is a prospective, interventional, randomized, open-label, controlled trial. It is supported by recent scholarly, peer-reviewed literature. The research method reflects the approach needed to answer the research questions. Research is addressing a gap in the literature that would contribute new findings. The research topic is based on a tangible and cited problem. The research collects and analyses the data, any deviations are documented and approved by NJUCM. The study was designed originally. The acupuncture treatment plan for KOA is designed with the assistance of Professor Xueping Zhou. The study will be conducted in a Family Medicine practice by the experimenter. All financial and operating burdens will be funded from practice resources.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Knee Osteoarthritis
* Knee Osteoarthritis for at least 6 months
* painful knee in last month
* radiographic changes of the knee (Kellgren-Lawrence grade 2 or more)
* signed informed consent
* participant can move independently

Exclusion Criteria:

* if the participant got knee intra-articular injection 3 months before his entry into the study
* uncontrolled malignant disease
* unstable heart disease
* advanced organ failure disease (NYHA III or IV, or a more than the twofold increase of creatinin, or marked dyspnea)
* unstable psychiatrist's disease
* bleeding diathesis
* anticoagulant use

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2022-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Svijetlana Perculija Durdevic, M.D., Principal Investigator — Family Medicine Practice Svijetlana Perculija Durdevic, MD
Locations (1):
- Family Medicine Practice Svijetlana Perculija Durdevic, MD, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlies the results reported in this article after deidentification (text, tables, figures, and appendices) for qualified researchers. Approval of the request is a prerequisite to the sharing of data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months following publication, ending 3 years following article publication
Access Criteria: Access to trial IPD can be requested by a qualified researcher engaging in independent scientific research.
  For more information or to submit a request please contact svijetlana.perculija.durdevic@outlook.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process was carried out from January 2021 to August 2021. The recruitment was performed at the Family Medicine practice, run by the investigator, who has access to the database of four thousand patients from two practices. From the 4000 patients, 180 made the target population by criteria ≥50 years and confirmed KOA from a computer database. A study population of 64 participants was made by applying the inclusion and exclusion criteria.
Pre-assignment Details: In the pre-assignment period, all 64 enrolled participants were assigned in a concealed manner to the A or C group.
Groups:
- Acupuncture Group: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to analgesics, whose dose could vary according to the participant's need. Participants and investigators were not blinded by treatment type, but assessors were blinded about the fact to which group participants belonged.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete treatment lasted 30 minutes.
  Conventional Medical Treatment: Participants took analgesics, prescribed by their general practitioner. They could modify the analgesics' dose according to the intensity of their symptoms.
- Control Group: 32 randomised participants allocated to the Control group got their standard conventional treatment (analgesics) whose dose varied according to the participant's symptoms intensity. Both participants and investigator were not blinded by treatment type. Assessors were blinded to the fact to which group participants belong.
  Conventional Medical Treatment: Participants took prescribed standard conventional medical treatment for pain or analgesics. Analgesics therapy was prescribed by their general practitioner. Participants modified the dose of analgesics according to the intensity of their symptoms.
Period: Week 1-24, Between Group Analysis
Arm/Group | Acupuncture Group | Control Group
Started (Start of acupuncture treatment of A group.) | 32 | 32
End of Acupuncture Treatments Treatment of A Group | 25 | 30
9 Weeks After Completing the Acupuncture Treatment | 25 | 29
Completed (Completion of the first study part at Week 24, 9 weeks after acupuncture treatment ended.) | 25 | 29
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 1 | 0
Period: Week 25-39, Within Group Analysis
Arm/Group | Acupuncture Group | Control Group
Started (Start of acupuncture treatments of C group (cross-over of C) at Week 25) | 25 | 29
Completed | 23 | 23
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Acupuncture Group: Participants in the Acupuncture (A) group got acupuncture treatments for their knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with a frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) whose dose varied according to participant symptoms intensity. The participants and investigator were not blinded by treatment type. The assessors were blinded for the fact to which group participants belong.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles were manipulated three times, every ten minutes, three times in total. The complete time of treatment was 30 minutes. All treatments were equally long.
  Conventional Medical Treatment: Participants took their standard conventional medical treatment (analgesics). Analgesics therapy was prescribed by their general practitioner. The participants modified the dose of analgesics according to the intensity of their symptoms.
- Control Group: Participants in the Control (C) group got their standard conventional treatment (analgesics) whose dose could vary according to the participants' symptoms intensity. Participants and investigator were not blinded for treatment type. The assessors were blinded for the fact to which group participants belong.
  Conventional Medical Treatment: Participants took their standard conventional medical treatment or analgesics. Analgesics therapy was prescribed by their general practitioner. The participants modified the dose of analgesics according to the intensity of their symptoms.
- Total: Total of all reporting groups
Arm/Group | Acupuncture Group | Control Group | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] — The average age of participants was 64 years, ranging from 50 to 81 years because the inclusion criteria for participant enrolment in the study was the age of 50 years or older.
  years | 64.1 (7.94) | 64.7 (8.27) | 64.4 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants] — The study sample of participants included 15 (23.4%) males and 49 (76.6%) females. Knee osteoarthritis occurs more often in females.
  Participants
    Female | 25 | 24 | 49
    Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — All participants from the study belong to the white race.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 32 | 32 | 64
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI), Continuous [Mean (Standard Deviation); unit: kg/m2] — Participants' average body mass index (BMI) in the study was 31.0 ( 31.4 in A and 30.6 in C group). The values of BMI range from 21,0 to 47,5 among participants. Obesity is one of the risk factors for knee osteoarthritis.
  kg/m2 | 31.4 (5.45) | 30.6 (5.70) | 31.0 (5.55)
Kellgren-Lawrence (K-L) grade, Categorical [Count of Participants; unit: Participants] — The average Kellgren-Lawrence (K-L) score was 3 in both groups, the scores range from 2 to 4 because a score of 2 was the minimum score for enrolling participants in the study. The grading of K-L participants could have shifted toward higher grades if the radiographs had been renewed before the start of the study. Existing patient recordings were used in the study. K-L grade was used here more for disease confirmation purposes.
  Participants
    grade 2 | 7 | 9 | 16
    grade 3 | 19 | 13 | 32
    grade 4 | 6 | 10 | 16
WOMAC total, Continuous [Mean (Standard Deviation); unit: score on a scale] — Western Ontario and McMaster University Osteoarthritis Index (WOMAC) is a renowned questionnaire used by health professionals to evaluate the condition of patients with KOA. It is an interval scale with a range from minimal 0 to maximal 96 points, a higher score supposes advanced osteoarthritis or a worse outcome and a lower score signifies better OA outcome presentation. It comprises 5 questions for pain (0-20), 2 for stiffness (0-8) and 17 for functional limitation (0-68) which all summed provide WOMAC total.
  score on a scale | 56.4 (18.908) | 57.3 (20.20) | 56.9 (19.414)
WOMAC pain, Continuous [Mean (Standard Deviation); unit: score on a scale] — Western Ontario and McMaster University Osteoarthritis (WOMAC) pain subscale of the WOMAC index evaluates OA pain by participants. It comprises 5 questions for pain assessed by a 5-point Likert scale between range from minimal 0 to maximal 20 points. A bigger score presents a worse outcome and a lower score relates to a better outcome.
  score on a scale | 11.5 (4.607) | 11.7 (4.37) | 11.6 (4.457)
WOMAC stiffness, Continuous [Mean (Standard Deviation); unit: score on a scale] — Western Ontario and McMaster University Osteoarthritis (WOMAC) stiffness subscale of the WOMAC index and evaluate knee OA stiffness by participants. It comprises 2 questions for stiffness assessed by a 5-point Likert scale between the range from minimal 0 to maximal 8 points. A bigger score presents a worse outcome and a lower score relates to a better result. WOMAC stiffness measures the stiffness of the knees.
  score on a scale | 3.8 (1.505) | 4.2 (2.20) | 4.0 (1.877)
WOMAC functional disability, Continuous [Mean (Standard Deviation); unit: score on a scale] — Western Ontario and McMaster University Osteoarthritis (WOMAC) functional disability subscale of the WOMAC index evaluates KOA functional disability by participants. It comprises 17 questions for functional disability assessed by a 5-point Likert scale between the range from minimal 0 to maximal 68 points. A bigger score presents a worse outcome and a lower score relates to a better result.WOMAC functional disability measures the functional disability of the knees.
  score on a scale | 40.8 (14.123) | 41.9 (14.88) | 41.5 (14.292)
VAS, Continuous [Median (Standard Deviation); unit: score on a scale] — VAS continuous scale of 100 mm in length is a widely used and recognized scale for pain intense assessment. The number of millimetres on the scale range from 0 to 100, where 0 represents no pain and 100 represents the maximal possible pain. The one millimetre represents one unit of scale. The scale was divided into 10 parts for easier quantifying knee pain by participants.
  score on a scale | 59.5 (22.767) | 59.1 (18.11) | 59.3 (20.41)
KDSQ, Continuous [Mean (Standard Deviation); unit: score on a scale] — The Kidney Deficiency Syndrome Questionnaire (KDSQ) is a valid reliable measure for the evaluation of KDS. Of all 39 symptoms of Kidney deficiency, the authors excluded symptoms related to childhood and the male gender. KDSQ represents a valid form for the evaluation of KDS for this sample when the question about vaginal dryness was excluded. KDSQ comprises 21 questions, which are evaluated in the form of a 4-point Likert scale, about various related symptoms and traits. The maximal score is 69, a higher score relates to a worse outcome, and a lower score signifies a better condition/outcome.
  score on a scale | 27.2 (11.105) | 26.2 (11.89) | 26.7 (11.427)
DRUG /IBU, Continuous [Mean (Standard Deviation); unit: milligram-equivalent of ibuprofen] — DRUG is an average daily dose of analgesics in the last three days before assessment, according to the statement of the participants; various kinds of analgesics used were recalculated in a comparable dose of the selected representative (ibuprofen), as the most prescribed one. DRUG is expressed in ibuprofen equivalent milligram units (IBU): various analgesic doses were converted into comparable doses of ibuprofen according to specified minimal, maximal, and medium daily analgesic doses, frequently used in daily clinical work. Baseline values range from 0 to 4400 mg IBU among participants.
  milligram-equivalent of ibuprofen | 637.5 (1095.960) | 625 (841.66) | 631.3 (969.352)
Active flexion L and R knees, Continuous [Mean (Standard Deviation); unit: degree of angle] — Knee active flexion is measured with a goniometer and expressed in degrees of angle (deg.). The maximal knee active flexion is 135 degrees, and the minimal is 0 degrees. A lower value represents a worse outcome, and a higher value represents a better outcome. Knee active flexion and knee active extension form the knee's range of movement. Population: Some participants did not respond to the measurement.
  degree of angle
    Active flexion L knee: number analyzed (Participants) | 29 | 30 | 59
    Active flexion L knee | 95.103 (17.707) | 89.167 (23.159) | 92.08 (20.70)
    Active flexion R knee: number analyzed (Participants) | 29 | 30 | 59
    Active flexion R knee | 93.448 (16.802) | 88.666 (21.573) | 91.02 (19.360)
Active extension L and R knee, Continuous [Mean (Standard Deviation); unit: degree of angle] — Knee active extension is measured with a goniometer and is expressed in degrees of angle (deg.). The normal range is from 0 to 5 degrees, where the reduced extension represents the flexion contracture. Possible values out of the range present knee laxity (if >5 degrees) or flexion contracture (if <0 degrees). Higher deviation represents worse outcomes, and lower deviation represents better outcomes. Values between 0 and 5 degrees are in the physiological range. Population: Some participants did not respond to the measurement.
  degree of angle
    Active extension L knee: number analyzed (Participants) | 29 | 30 | 59
    Active extension L knee | 0.586 (1.783) | 0.5 (1.526) | 0.54 (1.643)
    Active extension R knee: number analyzed (Participants) | 29 | 30 | 59
    Active extension R knee | 0.759 (2.370) | 0.5 (1.526) | 0.63 (1.973)
Circumference of L and R upper leg, Continuous [Mean (Standard Deviation); unit: centimeter] — The circumference of the thigh, at 15 centimetres above the patellar superior margin, by a measuring tape. It is an objective knee physical measure. The unit of measure is a centimetre (cm). In the observed periods, the measure estimates muscular strength or knee activity. Increased values indicate increased muscular strength/knee function (better outcomes), and decreased values indicate worse muscular strength /knee function (worse outcomes). Population: Some participants did not respond to the measurement.
  centimeter
    Circumference of L upper leg: number analyzed (Participants) | 29 | 30 | 59
    Circumference of L upper leg | 57.931 (5.941) | 55.607 (5.755) | 56.75 (5.914)
    Circumference of R upper leg: number analyzed (Participants) | 29 | 30 | 59
    Circumference of R upper leg | 58.121 (5.648) | 56.26 (5.613) | 57.17 (5.660)
Circumference of L and R knee, Continuous [Mean (Standard Deviation); unit: centimeter] — Circumference of the knee is an objective measure performed with a measuring tape. The unit of measure is a centimeter (cm). The knee could be enlarged due to obesity, inflammation and deformation (abnormal bone growth). Increased values indicate a higher level of knee inflammation /deformation and obesity. Population: Some participants did not respond to the measurement.
  centimeter
    Circumference of L knee: number analyzed (Participants) | 29 | 30 | 59
    Circumference of L knee | 42.610 (4.26) | 41.973 (3.279) | 42.29 (3.773)
    Circumference of R knee: number analyzed (Participants) | 29 | 30 | 59
    Circumference of R knee | 42.966 (4.598) | 42.013 (3.168) | 42.48 (3.931)

OUTCOME MEASURES:

1. Primary Outcome: WOMAC Total in Week 15
Description: The Western Ontario and McMaster University Osteoarthritis Index (WOMAC) total score is the sum of the three subscales: pain, stiffness, and functional disability.
  The minimum value is 0, and the maximum value is 96, where the lower score/value represents a better outcome, and the higher score/value represents a worse outcome.
Time Frame: Week 15
Population: WOMAC total in Week 15 estimates the immediate treatment effects of acupuncture on pain, stiffness and knee function when acupuncture treatments ended in a between-groups A and C analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- A Group in Week 15: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) which dose could vary according to the participant's symptoms intensity. Participants and investigators were not blinded by treatment type, but assessors were blinded by the fact to which group participants belong.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment was 30 minutes. All treatments were equally long.
  Conventional Medical Treatment: Participants took their standard conventional medical treatment (analgesics). Analgesics therapy was prescribed by their general practitioner. The participants modified the dose of analgesics according to the intensity of their symptoms.
- C Group in Week 15: 32 randomised participants allocated to the Control group got their standard conventional treatment (analgesics) whose dose varied according to the participant's symptoms intensity. Both participants and investigator were not blinded by treatment type. Assessors were blinded to the fact to which group participants belong.
  Conventional Medical Treatment: Participants took prescribed standard conventional medical treatment for pain or analgesics. Analgesics therapy was prescribed by their general practitioner. Participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 25 | 30
score on a scale | 11.6 (11.633) | 54.4 (19.4)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; WOMAC total analysis between groups at Week 15. The Shapiro-Wilk test (S-W) was used for testing the normality of the data distribution. The comparability of groups regarding specified variables to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -42.8 — mean (WOMAC total of group A in Week 15) - mean (WOMAC total of group C in Week 15)

2. Secondary Outcome: WOMAC Pain in Week 15
Description: Western Ontario and McMaster University Osteoarthritis (WOMAC) pain subscale, separated from the WOMAC index, evaluates knee OA pain by participants. It comprises 5 questions for pain assessed by a 5-point Likert scale ranging from minimal 0 to maximal 20 points. A bigger score presents a worse outcome, and a lower score relates to a better outcome.
Time Frame: Week 15
Population: WOMAC pain in Week 15 estimates the immediate treatment effects of acupuncture at Week 15 on knee OA pain after acupuncture treatments were completed in a between-groups A and C analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- C Group in Week 15: 32 randomized participants allocated to the Control group got their standard conventional treatment (analgesics) whose dose varied according to the participant's symptoms intensity. Both participants and investigator were not blinded by treatment type. Assessors were blinded to the fact to which group participants belong.
  Conventional Medical Treatment: Participants took prescribed standard conventional medical treatment for pain or analgesics. Analgesics therapy was prescribed by their general practitioner. Participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 25 | 30
score on a scale | 2.4 (2.4) | 11.3 (4.6)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; WOMAC pain analysis between groups at Week 15. The Shapiro-Wilk test (S-W) was used for testing the normality of the data distribution. The comparability of groups regarding specified variables to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at assessments; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -8.9 — mean (WOMAC pain of group A at Week 15) - mean (WOMAC pain of group C at Week 15)

3. Secondary Outcome: WOMAC Stiffness in Week 15
Description: Western Ontario and McMaster University Osteoarthritis (WOMAC) stiffness subscale, separated from the WOMAC index, and evaluate knee OA stiffness by participants. It comprises 2 questions for stiffness assessed by a 5-point Likert scale between the range from minimal 0 to maximal 8 points. A bigger score presents a worse outcome, and a lower score relates to a better result. WOMAC stiffness measures the stiffness of the knees.
Time Frame: Week 15
Population: WOMAC stiffness in Week 15 estimates the immediate treatment effects of acupuncture on knee OA stiffness after acupuncture treatments were completed at Week 15 in a between-groups A and C analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 25 | 30
score on a scale | 0.7 (0.9) | 4.6 (1.9)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; WOMAC stiffness between groups at Week 15. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups regarding specified variables to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -3.9 — mean (WOMAC stiffness of group A at Week 15) - mean (WOMAC stiffness of group C at Week 15)

4. Secondary Outcome: WOMAC Functional Disability in Week 15
Description: Western Ontario and McMaster University Osteoarthritis (WOMAC) functional disability subscale, separated from the WOMAC index, evaluates knee OA functional disability by participants' estimation. It comprises 17 items for functional disability assessment by a 5-point Likert scale ranging from minimal 0 to maximal 68 points. A bigger score presents a worse outcome, and a lower score relates to a better result. WOMAC functional disability measures climbing, rising from a chair/bed, standing, bending, walking, getting in/out of a car/bath/toilet, shopping, putting on socks, sitting and difficulties in domestic duties.
Time Frame: Week 15
Population: WOMAC functional disability in Week 15 estimates the immediate treatment effects of acupuncture on knee OA functional disability after acupuncture treatments were completed at Week 15 in a between-groups A and C analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 25 | 30
score on a scale | 8.6 (8.8) | 38.6 (13.9)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; WOMAC functional disability between groups at Week 15. The Shapiro-Wilk test (S-W) tests normality distribution. Furthermore, the comparability of groups regarding specified variables to accept or reject the null hypothesis of equality was tested with the Mann-Whitney U test, with a power of 95 % and a level of significance α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data at specified assessment (the mid-spread); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -30.0 — mean (WOMAC functional disability of group A in Week 15) - mean (WOMAC functional disability of group C in Week 15)

5. Secondary Outcome: VAS in Week 15
Description: Visual Analogue Scale (VAS) assesses knee OA pain intensity, ranging from 0 to 100; the lower value represents a better outcome, and the higher a worse outcome.
Time Frame: Week 15
Population: VAS 15 measure estimates the treatment effect of acupuncture on KOA pain at the acupuncture treatment completion time point, analysed between the A and C groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 25 | 30
score on a scale | 12.6 (12) | 61 (19.5)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; Visual Analogue Scale (VAS) was compared between groups at Week 15, when the acupuncture of group A ended. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) presented the statistical dispersion of sample data at specified assessments; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -48.4 — mean (VAS of group A in Week 15) - mean (VAS of group C in Week 15)

6. Secondary Outcome: KDSQ in Week 15
Description: The Kidney Deficiency Syndrome Questionnaire (KDSQ) assesses the intensity of Kidney deficiency (KD) symptoms; the minimum value is 0, and the maximum is 69. A lower score/value represents a better outcome, and a higher score/value represents a worse outcome.
  This measure represents the effect of acupuncture treatment on KD.
Time Frame: Week 15
Population: KDSQ in Week 15 estimates the treatment effect of acupuncture on Kidney deficiency symptoms at the end of the acupuncture treatments, analysed between the A and C groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 25 | 30
score on a scale | 10.8 (6.7) | 24.8 (12.5)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; The Kidney Deficiency Syndrome Questionnaire (KDSQ) was compared between groups in Week 15. The Shapiro-Wilk test (S-W) tests the normality of data distribution. The comparability of groups regarding the null hypothesis of similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were used to analyse the statistical dispersion of specified sample data at specified assessment; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -14.0 — mean (KDSQ of group A in Week 15) - mean (KDSQ of group C in Week 15)

7. Secondary Outcome: DRUG in Week 15
Description: DRUG is a measure that represents analgesics taken by participants, including various non-steroid anti-inflammatory drugs (NSAIDS) and/or tramadol. Recorded analgesics' doses from the last three days before assessment were recalculated in the comparable dose of the selective representative (ibuprofen) and converted into equivalent dose of milligrams of ibuprofen-ibuprofen equivalent units (IBU). DRUG's units of measure are IBU (units) on the scale ranging from 0 IBU to 4.500 IBU. DRUG decreasement represents a better therapeutic outcome, and an increase in DRUG represents a worse therapeutic outcome. All participants could self-manage the dosage according to their pain.
Time Frame: Week 15
Population: DRUG in Week 15 estimates the treatment effect of acupuncture on knee OA pain at the end of acupuncture treatment, analysed between groups A and C.
Measure: Mean (Standard Deviation); unit: milligrams-equivalent of ibuprofen(IBU)
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 25 | 30
milligrams-equivalent of ibuprofen(IBU) | 96.0 (183.7) | 870.0 (950.2)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; In Week 15, DRUG was compared between groups. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups regarding specified variables to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -774 — mean (DRUG of A group in Week 15) - mean (DRUG of C group in Week 15)

8. Secondary Outcome: Active Extension L and R Knees in Week 15
Description: The active extension of the left (L) and right (R) knees in Week 15 is an objective measure taken by an independent physiatrist with a goniometer, expressed on a scale with degrees of a goniometer angle as units.
  Knee active extension ranges between 0 and 5 degrees: the higher scores represent knee laxity/instability, and the negative scores represent knee flexion contraction. The higher values represent worse outcomes, and the lower values represent better outcomes.
Time Frame: Week 15
Population: Active extension of L and R knees in Week 15 represents the treatment effect of acupuncture on the knee OA at the completed acupuncture treatment time point in Week 15, compared between groups A and C.
Measure: Mean (Standard Deviation); unit: degrees of a goniometer angle
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 28 | 29
degrees of a goniometer angle
  L knee active extension | 0.429 (1.6) | 0.42 (1.35)
  R knee active extension | 0.607 (2.27) | 0.714 (1.78)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; Active extension of left (L) knees in Week 15 in the between-group analysis. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p = 0.8493, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.009 — mean (A group L knee in Week 15) - mean (C group L knee in Week 15)
Statistical Analysis 2: Comparison: A Group in Week 15 vs C Group in Week 15; Active extension of the right (R) knees in Week 15 in the between-group analysis. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p = 0.69654, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.107 — mean (A group R knee in Week 15) - mean (C group R knee in Week 15)

9. Secondary Outcome: Active Flexion L and R Knees in Week 15
Description: Active flexion of left (L) and right (R) knees in Week 15 is an objective measure provided by an independent physiatrist with a goniometer, expressed on a scale with degrees of a goniometer angle (units).
  Knee active flexion ranges from 0 to a maximum of 135 degrees; the lower score/value represents a worse outcome, and the higher score/value a better one.
Time Frame: Week 15
Population: Active flexion of L and R knees in Week 15 represents the treatment effect of acupuncture on knee function at the end of acupuncture treatment, Week 15, between groups A and C at Week 15.
Measure: Mean (Standard Deviation); unit: degrees on a goniometer angle
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 28 | 29
degrees on a goniometer angle
  L knee active flexion | 94.1 (17.1) | 90.2 (18.9)
  R knee active flexion | 96.1 (17.3) | 91.4 (18.6)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; L knee flexion between groups at Week 15. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p = 0.490, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3.9 — mean (active flexion L knee of group A at Week 15) - mean (active flexion L knee of group C at Week 15)
Statistical Analysis 2: Comparison: A Group in Week 15 vs C Group in Week 15; Right (R) knee flexion between groups in Week 15. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups regarding specified variables to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p = 0.517, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 4.7 — mean (active flexion R knee of group A at Week 15) - mean (active flexion R knee of group C at Week 15)

10. Secondary Outcome: Circumference of L and R Upper Leg in Week 15
Description: Circumference of the left (L) and right (R) upper leg in Week 15 is an objective measure, assessed by an independent physiatrist, at the thigh 15 centimetres above the patellar superior margin, measured with a tape measure. The unit of measure is a centimetre (unit) on the measuring tape (scale) with a range from 0 to 100 centimetres. This measure represents a measure of muscular strength or atrophy. Higher values indicate better outcomes from higher muscular volume, and decreased values indicate worse outcomes from weaker muscular volume.
Time Frame: Week15
Population: This measure estimates the treatment effect of acupuncture on knee function at the end of the acupuncture treatment time point in Week 15, in the between-groups A and C analysis.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 28 | 29
centimeters
  L upper leg circumference | 55.3 (5.84) | 58.3 (5.87)
  R upper leg circumference | 58.7 (6.88) | 55.7 (9.25)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; Circumference of the left (L) upper leg between groups analysis at Week 15. For group normality statistics, the Shapiro-Wilk test (S-W) was used. Furthermore, the comparability of groups regarding specified variables to accept or reject the hypothesis of equality was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of specified sample data at specified assessment; Test type: Superiority; p = 0.083, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -3.0 — mean (circumference of L upper leg of group A at Week 15) - mean (circumference of L upper leg of group C at Week 15)
Statistical Analysis 2: Comparison: A Group in Week 15 vs C Group in Week 15; Circumference of the right (R) upper leg between groups analysis at Week 15. For group normality statistics, the Shapiro-Wilk test (S-W) was used. Furthermore, the comparability of groups regarding specified variables to accept or reject the hypothesis of equality was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p = 0.084, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 3.0 — mean (circumference of R upper leg of group A at Week 15) - mean (circumference of R upper leg of group C at Week 15)

11. Secondary Outcome: Circumference of L and R Knees in Week 15
Description: Circumference of left (L) and right (R) knees at Week 15 is an objective measurement taken by an independent physiatrist; the measure includes the difference in circumference of the knees measured with a tape measure at the middle of the patellae. The unit of measure is a centimetre (unit) on the measuring tape (scale) with a range from 0 to 100 centimetres. This measure represents knee inflammation and joint deformation (abnormal bone growth). Increased values indicate worse outcomes from a higher level of knee inflammation/deformation, and decreased values indicate better outcomes from a lower level of knee inflammation/deformation.
Time Frame: Week 15
Population: Circumference of L and R knees in Week 15 estimates the treatment effect of acupuncture on knee osteoarthritis at the end of the acupuncture treatment time point, analysed between groups A and C.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | A Group in Week 15 | C Group in Week 15
Number analyzed (Participants) | 28 | 29
centimeters
  L knee circumference | 43.1 (3.9) | 41.8 (3.23)
  R knee circumference | 43.1 (4.14) | 41.8 (3.0)
Statistical Analysis 1: Comparison: A Group in Week 15 vs C Group in Week 15; Circumference of the left (L) knee in Week 15 was analysed between groups. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p = 0.341, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.3 — mean (circumference of L knee of group A at Week 15) - mean (circumference of L knee of group C at Week 15)
Statistical Analysis 2: Comparison: A Group in Week 15 vs C Group in Week 15; Circumference of the right (R) knee in between groups at Week 15. The Shapiro-Wilk test (S-W) was used to test the data distribution's normality. The comparability of groups to accept or reject the null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and standard deviation (SD) were calculated to present the statistical dispersion of sample data at specified assessments; Test type: Superiority; p = 0.317, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.3 — mean (circumference of R knee of group A at Week 15) - mean (circumference of R knee of group C at Week 15)

12. Secondary Outcome: WOMAC Total in Week 24
Description: Western Ontario and McMaster University Osteoarthritis (WOMAC) index's total score is a sum of all three subscales for pain, stiffness, and functional disability, the minimum value is 0, and the maximum value is 96; the lower score/value represents a better outcome, and a higher score/value represents a worse outcome
Time Frame: Week 24
Population: WOMAC total in Week 24 represents the treatment effect of acupuncture on pain, stiffness, and function at Assessment 9, in Week 24, nine weeks after acupuncture treatment ended, and was analysed between groups A and C.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- A Group in Week 24: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) which dose could vary according to the participant's symptoms intensity. Participants and investigators were not blinded by treatment type, but assessors were blinded by the fact to which group participants belong.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment was 30 minutes. All treatments were equally long.
  Conventional Medical Treatment: Participants took their standard conventional medical treatment (analgesics). Analgesics therapy was prescribed by their general practitioner. The participants modified the dose of analgesics according to the intensity of their symptoms.
- C Group in Week 24: 32 randomised participants allocated to the Control group got their standard conventional treatment (analgesics) whose dose varied according to the participant's symptoms intensity. Both participants and investigator were not blinded by treatment type. Assessors were blinded to the fact to which group participants belong.
  Conventional Medical Treatment: Participants took prescribed standard conventional medical treatment for pain or analgesics. Analgesics therapy was prescribed by their general practitioner. Participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 25 | 29
score on a scale | 20.4 (18.4) | 53.4 (20.5)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; WOMAC total was analysed in Week 24 between groups, nine weeks after acupuncture ended. The Shapiro-Wilk test (S-W) tested the normality of the distribution. The comparability of groups regarding specified variables to accept or reject the null hypothesis of equality was tested with the Mann-Whitney U test, with 95 % power and a level of significance α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of specified sample data at specified assessments; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -33.0 — mean (WOMAC total of group A in Week 24) -mean (WOMAC total of group C in Week 24)

13. Secondary Outcome: WOMAC Pain in Week 24
Description: Western Ontario and McMaster University Osteoarthritis (WOMAC) pain subscale, separated from the WOMAC index, evaluates OA pain by participants. It comprises 5 questions for pain assessed by a 5-point Likert scale, ranging from minimal 0 to maximal 20 points. A bigger score presents a worse outcome, and a lower score relates to a better one.
Time Frame: Week 24
Population: WOMAC pain in Week 24, nine weeks after acupuncture treatment ended, was analysed between groups A and C.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- C Group in Week 24: 32 randomized participants allocated to the Control group got their standard conventional treatment (analgesics) whose dose varied according to the participant's symptoms intensity. Both participants and investigator were not blinded by treatment type. Assessors were blinded to the fact to which group participants belong.
  Conventional Medical Treatment: Participants took prescribed standard conventional medical treatment for pain or analgesics. Analgesics therapy was prescribed by their general practitioner. Participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 25 | 29
score on a scale | 4.5 (3.7) | 11 (4.6)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; WOMAC pain was analysed between groups 9 weeks after acupuncture ended in Week 24. The Shapiro-Wilk test (S-W) tested the normality distribution. Furthermore, the comparability of groups regarding specified variables to accept or reject the hypothesis of equality was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of specified sample data (the mid-spread); Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -6.5 — mean (WOMAC pain of group A at Week 24) - mean (WOMAC pain of group C at Week 24)

14. Secondary Outcome: WOMAC Stiffness in Week 24
Description: Western Ontario and McMaster University Osteoarthritis (WOMAC) stiffness subscale, separated from the WOMAC index, evaluates knee OA stiffness by participants. It comprises 2 questions for stiffness assessed by a 5-point Likert scale ranging from minimal 0 to maximal 8 points. A bigger score represents a worse outcome, and a lower score relates to a better result. WOMAC stiffness measures the stiffness of the knees.
Time Frame: Week 24
Population: WOMAC stiffness in Week 24, nine weeks after acupuncture treatment ended, was analysed between groups A and C.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 25 | 29
score on a scale | 1.1 (1.5) | 3.4 (2.2)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; WOMAC stiffness between groups A and C in Week 24, 9 weeks after acupuncture ended. The Shapiro-Wilk test (S-W) tests the normality of distribution. Group comparability was tested with the Mann-Whitney U test with 95 % power and a level of significance α=0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of specified sample data at specified assessments; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -2.3 — mean (WOMAC stiffness of group A in Week 24) - mean (WOMAC stiffness of group C in Week 24)

15. Secondary Outcome: WOMAC Functional Disability in Week 24
Description: Western Ontario and McMaster University Osteoarthritis (WOMAC) functional disability subscale, separated from the WOMAC index, evaluates knee OA functional disability by participants' estimation. It comprises 17 items of functional disability assessment by a 5-point Likert scale ranging from minimal 0 to maximal 68 points. A bigger score presents a worse outcome, and a lower score relates to a better result. WOMAC functional disability measures climbing, rising from a chair/bed, standing, bending, walking, getting in/out of a car/bath/toilet, shopping, putting on socks, sitting, and difficulties in domestic duties.
Time Frame: Week 24
Population: WOMAC functional disability in Week 24 estimates the effects of acupuncture on functional disability nine weeks after the acupuncture treatment of knee OA ended, using a between-groups A and C analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 25 | 29
score on a scale | 14.7 (13.7) | 39.0 (14.5)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; WOMAC functional disability at Week 24 was analysed between groups. The Shapiro-Wilk test (S-W) tests the normality of data. The comparability of groups regarding specified variables (to accept or reject the null hypothesis of comparability) was tested with the Mann-Whitney U test with 95% power and a level of significance α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of specified sample data at specified assessments; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -24.3 — mean (WOMAC functional disability of group A in Week 24) - mean (WOMAC functional disability of group C in Week 24)

16. Secondary Outcome: VAS in Week 24
Description: as for outcome 5
Time Frame: Week 24
Population: VAS in Week 24 estimates the treatment effect of acupuncture on knee pain, 9 weeks after acupuncture treatment ended, in between groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 25 | 29
score on a scale | 13.8 (13.9) | 59.5 (23.9)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; VAS was compared between groups in Week 24. For group normality statistics, the Shapiro-Wilk test (S-W) was used. The comparability of groups regarding specified variables to accept or reject the hypothesis of equality was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -45.7 — mean (VAS in Week 24 of group A) - mean (VAS in Week 24 of group C)

17. Secondary Outcome: KDSQ in Week 24
Description: The Kidney Deficiency Syndrome Questionnaire (KDSQ) assesses the intensity of kidney deficiency symptoms; the minimum value is 0, and the maximum is 69. A lower score/value represents a better outcome, and a higher score/value represents a worse outcome.
  This measure represents the effect of acupuncture treatment on Kidney deficiency (KD).
Time Frame: Week 24
Population: KDSQ in Week 24 estimates the treatment effect of acupuncture on KD symptoms 9 weeks after acupuncture treatment ended, analysed between groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 25 | 29
score on a scale | 13.9 (8.9) | 25.0 (12.4)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; KDSQ between groups in Week 24. For group normality statistics, the Shapiro-Wilk test (S-W) was used. The comparability of groups regarding specified variables to accept or reject the hypothesis of equality was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -11.1 — mean (KDSQ in Week 24 of group A) - mean (KDSQ in Week 24 of group C)

18. Secondary Outcome: DRUG in Week 24
Description: as for outcome 7
Time Frame: Week 24
Population: DRUG in Week 24 estimates the treatment effect of acupuncture on knee OA pain nine weeks after the end of acupuncture treatment, analysed between groups A and C.
Measure: Mean (Standard Deviation); unit: milligrams-equivalent of ibuprofen(IBU)
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 25 | 29
milligrams-equivalent of ibuprofen(IBU) | 184.0 (395) | 765.5 (783)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; The DRUG between groups in Week 24. For group normality statistics, the Shapiro-Wilk test (S-W) was used. Furthermore, the comparability of groups regarding specified variables to accept or reject the hypothesis of equality was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -581.5 — mean (DRUG in Week 24 of group A) - mean (DRUG in Week 24 of group C)

19. Secondary Outcome: Active Extension L and R Knee in Week 24
Description: as for outcome 8
Time Frame: Week 24
Population: Active extension of L and R knee in Week 24 represents the treatment effect of acupuncture on the knee OA, nine weeks after the acupuncture treatment ended, compared between groups A and C.
Measure: Mean (Standard Deviation); unit: degrees of a goniometer angle
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 22 | 28
degrees of a goniometer angle
  Active extension of L knee at Week 24 | 0 (0) | 0 (0)
  Active extension of R knee at Week 24 | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; Left (L) knee analysis between groups A and C in Week 24. For group normality statistics, the Shapiro-Wilk test (S-W) was used. Furthermore, the comparability of groups regarding specified variables to accept or reject the hypothesis of comparability was tested with the Mann-Whitney U test, with 95% statistical power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data at assessment; Test type: Superiority; Mean Difference (Final Values) = 0.0 — mean (Act ext L of A group in Week 24) - mean (Act ext L of C group in Week 24)
Statistical Analysis 2: Comparison: A Group in Week 24 vs C Group in Week 24; Right (R) knee analysis between groups at Week 24. For group normality statistics, the Shapiro-Wilk test (S-W) was used. Furthermore, the comparability of groups regarding specified variables to accept or reject the hypothesis of comparability between groups was tested by the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data at specified assessment; Test type: Superiority; Mean Difference (Final Values) = 0.0 — mean (Act ext R knee of A group in Week 24) - mean (Act ext R knee of C group in Week 24)

20. Secondary Outcome: Active Flexion L and R Knees in Week 24
Description: as for outcome 9
Time Frame: Week 24
Population: Active flexion of L and R knees in Week 24 represents the treatment effect of acupuncture on knee function nine weeks after acupuncture treatment ended, compared between groups.
Measure: Mean (Standard Deviation); unit: degrees of a goniometer angle
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 22 | 28
degrees of a goniometer angle
  L knee | 98.6 (16.4) | 99.5 (24.8)
  R knee | 101.6 (22.1) | 99.8 (21.5)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; Left (L) knee flexion between groups at Week 24. The Shapiro-Wilk test (S-W) tests the normality of the distribution. Furthermore, the comparability of groups regarding specified variables to accept or reject the null hypothesis of equality was tested with the Mann-Whitney U test, with 95% power and a level of significance α = 0,05. Standard deviation (SD) was calculated to present the statistical dispersion of specified sample data at a specified assessment (time-point); Test type: Superiority; p = 0.953, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.9 — mean (L knee act flexion of group A in Week 24) - mean (L knee act flexion of group C in Week 24)
Statistical Analysis 2: Comparison: A Group in Week 24 vs C Group in Week 24; Right (R) knee flexion between groups at Week 24. The Shapiro-Wilk test (S-W) tests the normality of the distribution. Furthermore, the comparability of groups regarding specified variables to accept or reject the null hypothesis of comparability was tested with the Mann-Whitney U test, with 95% power and a level of significance α = 0,05. Standard deviation (SD) was calculated to present the statistical dispersion of sample data at an assessment; Test type: Superiority; p = 0.491, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.8 — mean (R knee act flexion of group A in Week 24) - mean (R knee act flexion of group C in Week 24)

21. Secondary Outcome: Circumference of L and R Upper Leg in Week 24
Description: Circumference of the left (L) and right (R) upper leg in Week 24 is an objective measure, assessed by an independent physiatrist, at the thigh 15 centimetres above the patellar superior margin, measured with a tape measure. The unit of measure is a centimetre (unit) on the measuring tape (scale) with a range from 0 to 100 centimetres. This measure represents a measure of muscular strength or atrophy. Higher values indicate better outcomes from higher muscular volume, and decreased values indicate worse outcomes from weaker muscular volume.
Time Frame: Week 24
Population: Circumference of L and R upper leg in Week 24 estimates the treatment effect of acupuncture on knee OA, nine weeks after the acupuncture treatment ended, analysed between groups.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 22 | 28
centimeters
  Circumference of L Upper Leg at Week 24 | 58.8 (5.59) | 57.2 (6.61)
  Circumference of R Upper Leg at Week 24 | 59.3 (5.93) | 57.2 (6.83)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; Circumference of the left (L) upper leg between groups in Week 24. The Shapiro-Wilk test (S-W) was used to test the normality of a distribution. The comparability of groups regarding specified variables to accept or reject the hypothesis of groups comparability was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data at assessments; Test type: Superiority; p = 0.261, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.6 — mean (circumference of L upper leg of group A in Week 24) - mean (circumference of L upper leg of group C in Week 24)
Statistical Analysis 2: Comparison: A Group in Week 24 vs C Group in Week 24; Circumference of the R upper leg between groups at Week 24. The Shapiro-Wilk test (S-W) was used to test the normality of distribution. The comparability of groups regarding specified variables (null hypothesis) was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range (IQR) and SD were analysed to present the statistical dispersion of sample data at assessments; Test type: Superiority; p = 0.273, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.1 — mean (circumference of R upper leg of group A in Week 24) - mean (circumference of R upper leg of group C in Week 24)

22. Secondary Outcome: Circumference of L and R Knee in Week 24
Description: as for outcome 21
Time Frame: Week 24
Population: Circumference of L and R Knee in Week 24 estimates the direct treatment effect of acupuncture on knee osteoarthritis, nine weeks after acupuncture treatment ended, analysed between groups.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- C Group in Week 24: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) which dose could vary according to the participant's symptoms intensity. Participants and investigators were not blinded by treatment type, but assessors were blinded by the fact to which group participants belong.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment was 30 minutes. All treatments were equally long.
  Conventional Medical Treatment: Participants took their standard conventional medical treatment (analgesics). Analgesics therapy was prescribed by their general practitioner. The participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 22 | 28
centimeters
  Circumference of L knees at Week 24 in between-groups | 43.6 (4.62) | 42.4 (4.14)
  Circumference of R knees at Week 24 in between-groups | 44.0 (4.38) | 42.4 (4.08)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; Circumference of left (L) knees in Week 24, in between-groups. The Shapiro-Wilk test (S-W) tests normality distribution. The comparability of groups regarding specified variables to accept or reject the null hypothesis of similarity was tested with the Mann-Whitney U test with 95% power and a level of significance α = 0,05. Standard deviation was calculated to present the statistical dispersion of sample data at an assessment; Test type: Superiority; p = 0.445, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.2 — mean (circumference of L knees in Week 24 of group A) - mean (circumference of L knees in Week 24 of group C)
Statistical Analysis 2: Comparison: A Group in Week 24 vs C Group in Week 24; Circumference of right (R) knees at Week 24 was analysed between groups. The Shapiro-Wilk test (S-W) tests normality distribution. The comparability of groups regarding specified variables to accept or reject the null hypothesis of similarity was tested with the Mann-Whitney U test with 95% power and a level of significance α = 0,05. Standard deviation was calculated to present the statistical dispersion of sample data at assessments; Test type: Superiority; p = 0.260, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.6 — mean (circumference of R knees in Week 24 of group A) - mean (circumference of R knees in Week 24 of group C)

23. Secondary Outcome: WOMAC Total in Week 39
Description: Western Ontario and McMaster University Osteoarthritis (WOMAC) total at the Added assessment at Week 39 in the crossover part compared to pre-experimental baseline value. The total score is a sum of all three subscales: pain, stiffness, and functional limitation. The minimum value is 0, and the maximum value is 96, where the lower score/value represents a better outcome, and a higher score/value represents a worse outcome.
Time Frame: Week 39
Population: WOMAC total in Week 39 represents the treatment effect of acupuncture on knee pain, stiffness, and function at the added assessment in Week 39 in the A and C groups compared to their baseline values by within-group analysis. It presents two: the magnitude of persisted effects 24 weeks after acupuncture treatment ended in group A, and the immediate effects of acupuncture treatment in group C in comparison with their baseline values.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- A Group in Week 39; A Group in Week 0: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) which dose could vary according to the participant's symptoms intensity. Participants and investigators were not blinded by treatment type, but assessors were blinded by the fact to which group participants belong.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment was 30 minutes. All treatments were equally long.
  Conventional Medical Treatment: Participants took their standard conventional medical treatment (analgesics). Analgesics therapy was prescribed by their general practitioner. The participants modified the dose of analgesics according to the intensity of their symptoms.
- C Group in Week 39; C Group in Week 0: 32 randomised participants allocated to the Control group got their standard conventional treatment (analgesics) whose dose varied according to the participant's symptoms intensity. Both participants and investigator were not blinded by treatment type. Assessors were blinded to the fact to which group participants belong.
  Conventional Medical Treatment: Participants took prescribed standard conventional medical treatment for pain or analgesics. Analgesics therapy was prescribed by their general practitioner. Participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | A Group in Week 39 | C Group in Week 39 | A Group in Week 0 | C Group in Week 0
Number analyzed (Participants) | 23 | 23 | 32 | 32
score on a scale | 22.0 (20.7) | 18.2 (17.62) | 56.4 (18.91) | 57.3 (20.2)
Statistical Analysis 1: Comparison: A Group in Week 39 vs A Group in Week 0; Western Ontario and McMaster University Osteoarthritis Index (WOMAC) total of group A in Week 39 (24 weeks after acupunctures ended) was compared with the pre-experimental baseline assessment by within-group analysis. The Shapiro-Wilk test (S-W) tests normality distribution. The null hypothesis at weeks 0 and 39 was tested with the Mann-Whitney U test with 95 % power and a level of significance α=0,05. Standard deviation (SD) was calculated to present the statistical dispersion of the sample; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -34.4 — mean (WOMAC total of group A in Week 39) - mean (WOMAC total of group A in Week 0)
Statistical Analysis 2: Comparison: C Group in Week 39 vs C Group in Week 0; WOMAC total of group C in Week 39 was tested for the significance level and mean difference by within-group analysis. The Shapiro-Wilk test (S-W) tests normality distribution. WOMAC total at Week 0 (pre-experimental baseline assessment) and Week 39 were compared to test the null hypothesis of group comparability by the Mann-Whitney U test with 95 % power and a level of significance α=0,05. Standard deviation (SD) was calculated to present the statistical dispersion of a sample; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -39.1 — mean (WOMAC total in Week 39 of group C) - mean (WOMAC total in Week 0 of group C)

24. Secondary Outcome: WOMAC Pain in Week 39
Description: The Western Ontario and McMaster University Osteoarthritis (WOMAC) pain subscale, selected from the WOMAC index, evaluates knee OA pain by participants. It comprises 5 questions for pain assessed by a 5-point Likert scale, ranging from minimal 0 to maximal 20 points. A bigger score presents a worse outcome, and a lower score relates to a better one.
Time Frame: Week 39
Population: WOMAC pain subscale in Week 39 by within-group analysis presented the magnitude of persisted pain reduction in group A (24 weeks after acupuncture treatment ended), and in group C, the immediate effects, when group C received acupuncture treatments after crossover in Week 25.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- A Group in Week 39; A Group in Week 0: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to analgesics, whose dose could vary according to the participant's need. Participants and investigators were not blinded by treatment type, but assessors were blinded about the fact to which group participants belonged.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete treatment lasted 30 minutes.
  Conventional Medical Treatment: Participants took analgesics, prescribed by their general practitioner. They could modify the analgesics' dose according to the intensity of their symptoms.
Arm/Group | A Group in Week 39 | C Group in Week 39 | A Group in Week 0 | C Group in Week 0
Number analyzed (Participants) | 23 | 23 | 32 | 32
score on a scale | 5.3 (4.72) | 4.7 (3.77) | 11.5 (4.61) | 11.7 (4.37)
Statistical Analysis 1: Comparison: A Group in Week 39 vs A Group in Week 0; The pain subscale of the WOMAC index of group A in Week 39 (24 weeks after acupunctures ended) was compared with baseline by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range and standard deviation were calculated to present the statistical dispersion of sample data at assessments; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -6.2 — mean (WOMAC pain in Week 39 of group A) - mean (WOMAC pain in Week 0 of group A)
Statistical Analysis 2: Comparison: C Group in Week 39 vs C Group in Week 0; The pain subscale of the WOMAC index of group C in Week 39 (end of acupuncture of group C) was compared with the pre-experimental baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range and standard deviation were calculated to present the statistical dispersion of data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -7.0 — mean (WOMAC pain in Week 39 of group C) - mean (WOMAC pain in Week 0 of group C)

25. Secondary Outcome: WOMAC Stiffness in Week 39
Description: as for outcome 14
Time Frame: Week 39
Population: WOMAC stiffness in Week 39 presents in group A the magnitude of persisted acupuncture effects 24 weeks after acupuncture treatment ended, and in group C, the immediate effects of acupuncture after group C crossed over in Week 25, analysed within-groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 39 | C Group in Week 39 | A Group in Week 0 | C Group in Week 0
Number analyzed (Participants) | 23 | 23 | 32 | 32
score on a scale | 1.2 (2.17) | 1.2 (1.95) | 3.8 (1.51) | 4.2 (2.20)
Statistical Analysis 1: Comparison: A Group in Week 39 vs A Group in Week 0; The stiffness subscale of the WOMAC index of group A in Week 39 (24 weeks after acupuncture of group A ended) was compared with the pre-experimental baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -2.6 — mean (WOMAC stiffness in Week 39 of group A) - mean (WOMAC stiffness in Week 0 of group A)
Statistical Analysis 2: Comparison: C Group in Week 39 vs C Group in Week 0; The stiffness subscale of the WOMAC index of group C in Week 39 (end of acupuncture of group C) was compared with the pre-experimental baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α = 0,05. Interquartile range and standard deviation were calculated to present the statistical dispersion of data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -3.0 — mean (WOMAC stiffness in Week 39 of group C) - mean (WOMAC stiffness in Week 0 of group C)

26. Secondary Outcome: WOMAC Functional Disability in Week 39
Description: as for outcome 4
Time Frame: Week 39
Population: WOMAC functional disability in Week 39 represents the treatment effect of acupuncture on knee functional disability at the added assessment in Week 39 in the A and C groups compared to their baseline values by within-group analysis. It presents two: the magnitude of persisted effects 24 weeks after acupuncture treatment ended in group A, and the immediate effects of acupuncture treatment in group C in comparison with their baseline values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 39 | C Group in Week 39 | A Group in Week 0 | C Group in Week 0
Number analyzed (Participants) | 23 | 23 | 32 | 32
score on a scale | 15.5 (14.3) | 12.3 (12.83) | 40.8 (14.12) | 41.9 (14.88)
Statistical Analysis 1: Comparison: A Group in Week 39 vs A Group in Week 0; The functional disability subscale of the WOMAC index of group A in Week 39 (24 weeks after acupuncture of group A ended) was compared with baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -25.3 — mean (WOMAC functional disability in Week 39 of group A) - mean(WOMAC functional disability in Week 0 of group A)
Statistical Analysis 2: Comparison: C Group in Week 39 vs C Group in Week 0; The functional disability subscale of the WOMAC index of group C in Week 39 (when acupuncture of group A ended) was compared with baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -29.6 — mean (WOMAC functional disability in Week 39 of group C) - mean (WOMAC functional disability in Week 0 of group C)

27. Secondary Outcome: VAS in Week 39
Description: Visual Analogue Scale (VAS) assesses knee OA pain intensity, ranging from 0 to 100; the lower value represents a better outcome, and the higher a worse outcome.
  This measure estimates the treatment effect of acupuncture on knee pain in Week 39 separately for groups A and C.
Time Frame: Week 39
Population: VAS in Week 39 presented two: group A was analysed for the magnitude of the persisted acupuncture effects 24 weeks after acupuncture ended, and the immediate acupuncture effect on knee pain was presented in group C.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- A Group in Week 39; A Group in Week 0: Participants in Acupuncture group will get acupuncture treatments to their symptomatic knee/knees according to the study protocol. Acupuncture will be provided to participants in three cycles, each three weeks duration, with frequency three times weekly. Period between the cycles is three weeks long. Participants will get acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) which dose could vary according to participant symptoms intensity. Participants and investigator are not blinded for treatment type.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment is 30 minutes. All treatments will be equal.
  Conventional Medical Treatment: Participants could take their standard conventional medical treatment or analgesics. Analgesics therapy is prescribed by their general practitioner. The dose of analgesics could be modified according to participants' symptoms intensity.
- C Group in Week 39: Participants in Control group will get their standard conventional treatment (analgesics) which dose could vary according to participant symptoms intensity. Participants and investigator are not blinded for treatment type.
  Conventional Medical Treatment: Participants could take their standard conventional medical treatment or analgesics. Analgesics therapy is prescribed by their general practitioner. The dose of analgesics could be modified according to participants' symptoms intensity.
- C Group in Week 0: Participants in the Control group will get their standard conventional treatment (analgesics) whose dose could vary according to the participant's symptoms intensity. Participants and investigator are not blinded by treatment type.
  Conventional Medical Treatment: Participants could take their standard medical treatment or analgesics. Analgesics therapy is prescribed by the general practitioner. The dose of analgesics could be modified according to participants' symptoms intensity.
Arm/Group | A Group in Week 39 | C Group in Week 39 | A Group in Week 0 | C Group in Week 0
Number analyzed (Participants) | 23 | 23 | 32 | 32
score on a scale | 18.3 (22.59) | 28.0 (21.36) | 59.5 (22.77) | 59.1 (18.1)
Statistical Analysis 1: Comparison: A Group in Week 39 vs A Group in Week 0; VAS of group A in Week 39 (24 weeks after acupuncture of group A ended) was compared with baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -41.2 — mean (VAS in Week 39 of group A) - mean (VAS in Week 0 of group A)
Statistical Analysis 2: Comparison: C Group in Week 39 vs C Group in Week 0; VAS of group C in Week 39 (when acupuncture of group C ended) was compared with baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -31.1 — mean (VAS in Week 39 of group C) - mean (VAS in Week 0 of group C)

28. Secondary Outcome: KDSQ in Week 39
Description: The Kidney Deficiency Syndrome Questionnaire (KDSQ) assesses the intensity of Kidney deficiency symptoms; the minimum value is 0, and the maximum is 69. A lower score/value represents a better outcome, and a higher score/value represents a worse outcome.
  This outcome represents the treatment effect of acupuncture on Kidney deficiency symptoms for both groups separately.
Time Frame: Week 39
Population: KDSQ in Week 39 represents the treatment effect of acupuncture on Kidney deficiency symptoms intensity at the completed acupuncture treatments time point in group C and the magnitude of persisted effects 24 weeks after acupuncture treatments ended in group A, compared with Week 0 by within-group analysis separately for both groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- A Group in Week 0: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) whose dose could vary according to the participant's symptoms intensity. Participants and investigators were not blinded by treatment type, but assessors were blinded by the fact to which group participants belong.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment was 30 minutes. All treatments were equally long.
  Conventional Medical Treatment: Participants took their standard medical treatment (analgesics). Their general practitioner prescribed analgesic therapy. The participants modified the dose of analgesics according to the intensity of their symptoms.
- C Group in Week 0: 32 randomised participants allocated to the Control group got their standard conventional treatment (analgesics) whose dose varied according to the participant's symptoms intensity. Both participants and investigator were not blinded by treatment type. Assessors were blinded to the fact to which group participants belonged.
  Conventional Medical Treatment: Participants took prescribed standard medical treatment for pain or analgesics. Their general practitioner prescribed analgesic therapy. Participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | A Group in Week 39 | C Group in Week 39 | A Group in Week 0 | C Group in Week 0
Number analyzed (Participants) | 23 | 23 | 32 | 32
score on a scale | 14.6 (9.12) | 14.8 (8.92) | 27.2 (11.10) | 26.2 (11.89)
Statistical Analysis 1: Comparison: A Group in Week 39 vs A Group in Week 0; KDSQ of group A in Week 39 (24 weeks after acupuncture of group A ended) was compared with baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -12.6 — mean (KDSQ in Week 39 of group A) - mean (KDSQ in Week 0 of group A)
Statistical Analysis 2: Comparison: C Group in Week 39 vs C Group in Week 0; KDSQ of group C in Week 39 (when acupuncture of group C ended) was compared with baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -11.4 — mean (KDSQ in Week 39 of group C) - mean (KDSQ in Week 0 of group C)

29. Secondary Outcome: DRUG by Added Assessment in Week 39, Crossover Part
Description: as for outcome 7
Time Frame: Week 39
Population: DRUG in Week 39 estimates the treatment effect of acupuncture on knee OA pain at the end of acupuncture treatment, analysed within groups A and C to present the effects of the 24-week period after acupuncture ended in group A, and the immediate effects in group C.
Measure: Mean (Standard Deviation); unit: milligrams-equivalent of ibuprofen(IBU)
Groups:
- A Group in Week 0: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) whose dose could vary according to the participant's symptoms intensity. Participants and investigators were not blinded by treatment type, but assessors were blinded by the fact to which group participants belong.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment was 30 minutes. All treatments were equally long.
  Conventional Medical Treatment: Participants took their standard medical treatment (analgesics). Their general practitioner prescribed analgesic therapy. The participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | A Group in Week 39 | C Group in Week 39 | A Group in Week 0 | C Group in Week 0
Number analyzed (Participants) | 23 | 23 | 32 | 32
milligrams-equivalent of ibuprofen(IBU) | 276.1 (566.46) | 319.6 (473.08) | 637.5 (1095.96) | 625.0 (841.66)
Statistical Analysis 1: Comparison: A Group in Week 39 vs A Group in Week 0; The DRUG of group A in Week 39 (24 weeks after acupuncture of group A ended) was compared with baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p = 0.204, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -361.4 — mean (DRUG in Week 39 of group A) - mean (DRUG in Week 0 of group A)
Statistical Analysis 2: Comparison: C Group in Week 39 vs C Group in Week 0; The DRUG of group C in Week 39 (when acupuncture of group C ended) was compared with baseline values by within-group analysis. The Shapiro-Wilk test (S-W) was used for testing the normality of the distribution. The null hypothesis of groups' similarity was tested with the Mann-Whitney U test, with 95% power and a significance level α=0,05. Interquartile range and SD were calculated to present the statistical dispersion of the data; Test type: Superiority; p = 0.134, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -305.4 — mean (DRUG in Week 39 of group C) - mean (DRUG in Week 0 of group C)

30. Secondary Outcome: Lequesne Index in Week 24, Between-group Analysis
Description: The Lequesne index is an algofunctional index of knee osteoarthritis that comprises three sections. Its score ranges from a minimal 0 (no pain and disability) to 24 (the greatest pain and disability). This index is added to the study in Week 24 as an additional objective measure. It measures pain severity with 5 questions, walking distance with 2 questions, and activities of daily living with 4 questions.
Time Frame: Week 24
Population: Groups A and C were compared in Week 24 using a between-groups analysis to assess the effect of the acupuncture treatment on Group A, as Group C served as the control up to Week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A Group in Week 24 | C Group in Week 24
Number analyzed (Participants) | 25 | 29
score on a scale | 5.1 (3.45) | 12.63 (5.06)
Statistical Analysis 1: Comparison: A Group in Week 24 vs C Group in Week 24; The Lequesne index in Week 24 compared two confirmed comparable groups (at baseline), 9 weeks after acupuncture treatment in group A ended, while the C group was still a control. The Shapiro-Wilk test (S-W) tests normality distribution. The between-group comparability test at Week 24 was provided to accept or reject the null hypothesis by the Mann-Whitney U test, with 95 % power and a level of significance α = 0,05. Standard deviation (SD) was calculated to present the statistical dispersion; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -7.53 — mean (Lequesne index in Week 24 of A group) - mean (Lequesne index in Week 24 of C group)

ADVERSE EVENTS:
Time Frame: The whole experiment lasted 39 weeks. The treatment protocol for every participant lasted 15 weeks. The treatment protocol comprises 3 cycles 3 weeks long, and between two cycles was a 3-week break. Participants could participate in 27 acupuncture sessions for 15 weeks in 3-times-weekly rhythm.
Description: Every participant had his own form for adverse events where the observer fulfilled adverse events.
Groups:
- Acupuncture Group: 32 randomised participants were allocated to the Acupuncture group to get acupuncture treatments for both knees according to the study protocol. Acupuncture was provided to participants in three cycles, each three weeks long, with the frequency of three times weekly. The period between the cycles was three weeks long. Participants got acupuncture as adjunctive therapy to conventional medical treatment (analgesic therapy) which dose could vary according to the participant's symptoms intensity. Participants and investigators were not blinded by treatment type, but assessors were blinded by the fact to which group participants belong.
  Acupuncture: Acupuncture treatment includes pricking the skin with acupuncture needles 0.3 x 40 millimetres in size, in the places of prescribed acupuncture points. Placed needles should be manipulated three times, every ten minutes, three times in total. The complete time of treatment was 30 minutes. All treatments were equally long.
  Conventional Medical Treatment: Participants took their standard conventional medical treatment (analgesics). Analgesics therapy was prescribed by their general practitioner. The participants modified the dose of analgesics according to the intensity of their symptoms.
Arm/Group | Acupuncture Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 2/32 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupuncture Group (N=32) | Control Group (N=32)
suprapatellar knee jount effusion (M13.1) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — at suprapatellar region effusion happened after treatment on the pace of pricking the skin, the change subsided within a few days
hematoma subcutaneus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — in the suprapubic region, subcutaneous bleeding happened with induration 4 cm in diameter, the change subsided in 10 days, directly related to pricking the skin with a needle
hematoma of upper leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — bruising suprapatellar 3-4 cm in diameter happened, was resolved in a 7 days

LIMITATIONS AND CAVEATS:
The assessor who did the physiatrist measurement was sick during 3rd assessment and because of that 3rd measurement, which differs in both groups from the previous two, was done with another assessor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT05014542/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT05014542/SAP_001.pdf
  • Informed Consent Form (2022-12-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT05014542/ICF_002.pdf